CLINICAL TRIAL: NCT01904188
Title: Clinical Microbial Species and Antibiotic Resistance Identification in Patients Presenting to the Emergency Department With Three of Four Systemic Inflammatory Response Syndrome (SIRS) Criteria - is Rapid Identification Possible and Accurate?
Brief Title: Clinical Microbial Species & Antibiotic Resistance ID in ED Patients Presenting With Infection - is Rapid ID Possible & Accurate?
Status: Recruiting | Type: Observational
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Mary Hughes, Professor of Emergency Medicine, Chair Department of Osteopathic Medical Specialties, Michigan State University
Other Study IDs: C13-033F
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Sepsis; Systemic Inflammatory Response Syndrome; Infection Mixed; Infection, Bacterial; Infection, Fungal; Infection, Coronavirus
Keywords: microbial identification; antibiotic resistance; In-Dx and other methods as developed; sepsis; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome; Coinfection; Bacterial Infections; Mycoses; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Prior to being analyzed the specimens will be retained in frozen state until there is a large enough quantity to batch run specimens in our investigational lab.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SIRS positive: Adult (> or = 18 years) patients with 3 of 4 systemic inflammatory response syndrome (SIRS) characteristics (1. tachycardia, 2. fever or hypothermia, 3. tachypnea, 4. leukocytosis), who have blood cultures drawn and urine collected for the evaluation of suspected sepsis, or those with a source of infection in any other bodily fluid suspected to be the source of infection. May also include others without SIRS criteria but with bodily fluid production or infection of a bodily fluid
  Interventions: Device: Gene Z or other rapid diagnostic techniques developed in our lab (as of 2018 not using Gene Z - now using In-Dx along with other developed techniquesregularly)

INTERVENTIONS:
Device: Gene Z or other rapid diagnostic techniques developed in our lab (as of 2018 not using Gene Z - now using In-Dx along with other developed techniquesregularly) — The Gene Z device (no longer in use) and now using In-Dx created in our lab, and other rapid diagnostic techniques that we have developed in our lab will be used to analyze previously processed specimens for microbial organisms and compared to prior culture and sensitivity results. It is not a separate arm - all samples will be cultured in lab per standard protocol and then the Gene Z device or other rapid diagnostic techniques developed in our lab will be used to re-analyze at a later date specimens that were previously frozen and stored and compared to culture results

SUMMARY:
The aim of this project is to test the utility of The Gene Z device (as of 2018 Gene Z no longer being used), now using In-Dx and other rapid identification techniques that the investigators have developed in the lab on clinically obtained bodily fluid samples taken from patients with suspected infection or sepsis based on having three of four positive Systemic Inflammatory Response Syndrome markers, or having a known infection for which a specimen is being collected. Specimens will be collected by University of Michigan Health/Sparrow Laboratories and McLaren Greater Lansing laboratories, processed and stored for analysis at a later date to determine if the microbial pathogens identified by current methods of culture, as well as pathogen susceptibility to antibiotics by culture results, can be identified by the GeneZ technology (no longer in use) or other developed technology accurately, and more timely. It will not affect current patient care nor impact patient care, which will continue in the standard fashion today for sepsis. Results will be compared to standard culture results and antibiotic sensitivities.

DETAILED DESCRIPTION:
Dramatic improvement in the timely and effective treatment of patients afflicted with sepsis can be achieved with the implementation of modern technologies for identification of offending microbial species and their innate genetic antibiotic treatment targets. Our collaborative team is planning to address this need using a Point-of-Care (POC) device equipped for identification of a bacterial species within 60 minutes of a routine Emergency Department laboratory blood draw or other specimen collection, followed by targeted analysis of its innate genetic antibiotic resistance elements within as little as 7 hours time. This revolutionary improvement in clinical management is critical for improving patient outcomes for a disease syndrome that is not only highly prevalent worldwide, consuming a massive amount of medical resources daily, but that only threatens to continue to worsen given current antibiotic stewardship practices. Early goal-directed therapy (EGDT) is the standard by which medical interventions are now shaped across fields in the modern clinical setting, ranging from trauma and neurosurgery to cardiology and infectious disease. Rapid and accurate diagnoses, paired with aggressive and effective intervention, are manifest to stemming the disease process as well as maintaining economically feasible care and improving long-term morbidity. The effort to apply EGDT to patients at high risk for systemic infection, sepsis, was initiated over a decade ago by Rivers and colleagues in the Emergency Department setting. Systematic approaches to early sepsis identification and intervention including broad-spectrum antibiotic coverage, and adequate fluid volume resuscitation have yielded definite improvements in patient outcomes and health care resource utilization. It has been recognized that one of the limiting factors in treatment of sepsis in the hospital setting is the timeliness of pathogen identification and implementation of appropriate antimicrobial therapy. The current "gold standard" of sepsis microbial identification is blood culture, which takes 3-5 days for a definitive species identification. Antimicrobial agent susceptibility for the given organism is generally garnered within this same time frame. However, in the period it takes from specimen collection to culture results, empiric broad-spectrum antibiotic coverage, often involving multiple antibiotics, must be provided to ensure organism eradication. This proposal aims to use Point of Care (POC) testing, as described by the investigatos' laboratory, to accurately identify pathogenic microorganisms in patients with suspected sepsis within 20 minutes of a laboratory blood draw or urine collection. The scope of the investigators' proposal is feasible in that 20 organisms account for 87% of microbial infections identified by culture-based techniques at University of Michigan Health/Sparrow Hospital, representing the greater Lansing, Michigan area, and 50 microorganisms would account for virtually every microbial infectious species (Khalife, 2011, unpublished data). In preliminary studies the investigators have validated this approach with laboratory-processed samples of Escherichia coli and Staphylococcus aureus. The investigators now are creating panels for multiple types of infections and have validated these efforts on over 30 microorganisms. POC testing will now be expanded to include additional microorganisms commonly encountered in sepsis patients or those with other identifiable infectious sources. Secondarily, antimicrobial resistance genes will be scanned using a functional genomics approach with highly-parallel quantitative PCR as performed by the investigators' laboratory in a previous study exploring the microbiota of porcine gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with 3 of 4 systemic inflammatory response syndrome (SIRS) characteristics (1. tachycardia, 2. fever or hypothermia, 3. tachypnea, 4. leukocytosis), who have blood cultures drawn and urine collected for the evaluation of suspected sepsis, and/or other bodily fluids collected for culture and sensitivity analysis.

Patients with other sources of infection with less than 3 of 4 SIRS criteria

Exclusion Criteria:

Pediatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who undergo evaluation for suspected sepsis who have peripheral blood cultures and urine samples obtained and patient characteristics recorded. In addition those that have an obvious infection without sepsis will be consented. Those that have other bodily fluids involved in addition will also be included, with or without SIRS criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2015-06; Primary Completion 2030-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of microbial identification with culture results from clinical laboratory | up to six months per specimen
  Frozen microbial specimens will be transported to an off site laboratory for analysis with the GeneZ or other point of care or rapid diagnostic technique or device, with investigators blinded to the final culture results of the specimen - positive or negative. Comparison will be made between final culture result and GeneZ identification of organism or other method as developed in the investigators' lab.

SECONDARY OUTCOMES:
Microbial Resistance Gene Pattern | up to one year per specimen
  Frozen specimens will be transported to an offsite laboratory where real time PCR will be used to identify microorganism resistance gene patterns of organisms identified by the GeneZ device or other rapid diagnostic technique or point of care device. These will be compared to the antibiotic sensitivity results from the culture and sensitivity reports done in the clinical laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Hughes, DO, Principal Investigator — Michigan State University
Locations (2):
- United States (2):
  - University of Michigan Health/Sparrow (name change only), Lansing, Michigan
  - McLaren Greater Lansing, Lansing, Michigan